CLINICAL TRIAL: NCT03036462
Title: Ferric Carboxymaltose Assessment of Morbidity and Mortality in Patients With IRon Deficiency and Chronic Heart Failure
Brief Title: Intravenous Iron in Patients With Systolic Heart Failure and Iron Deficiency to Improve Morbidity & Mortality
Acronym: FAIR-HF2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FAIR-HF2; FAIR-HF2-DZHK5 (Other Grant/Funding Number: Deutsches Zentrum für Herzkreislaufforschung)
Record Dates: First submitted 2016-09-15; First posted 2017-01-30 (Estimated); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Systolic Heart Failure; Iron Deficiency
Keywords: intravenous iron; systolic heart failure; iron deficiency; morbidity; mortality
MeSH Terms: conditions — Heart Failure, Systolic; Iron Deficiencies | interventions — Iron; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Verum group (FCM) (Experimental): I.v. iron administration in the form of FCM will be carried out according to SmPC. I.v. iron bolus administration (1000 mg) will be followed by an optional administration of 500-1000 mg within the first 4 weeks, (up to a total of 2000 mg which is in-label), according to the approved dosing rules, followed by administration of 500 mg FCM at every 4 months, except when haemoglobin is > 16.0 g/dL or ferritin is > 800 µg/L .In the verum group, all patients will receive a saline administration, when no iron is indicated at the time of the visit and according to the values listed above.
  Interventions: Drug: Iron
- Placebo group (NaCL) (Placebo Comparator): Administration of i.v. NaCl at a volume according to the dosing rules for FCM, i.e. as described for the verum group.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Iron — i.v. iron administration
  Arms: Verum group (FCM)
Drug: Saline — i.v. NaCl administration
  Other Names: salin
  Arms: Placebo group (NaCL)

SUMMARY:
The purpose of this study is to determine whether intravenous iron supplementation using ferric carboxymaltosis (FCM) extends the time-to-first-event of heart failure hospitalisations and cardiovascular (CV) death and reduces hospitalisation and mortality in patients with iron deficiency and heart failure.

DETAILED DESCRIPTION:
The clinical trial is designed as an international, prospective, multi-centre, double-blind, parallel group, randomised, controlled, interventional trial to investigate whether a long-term therapy with i.v. iron (ferric carboxymaltosis) compared to placebo can extend the time-to-first-event of heart failure hospitalisations and cardiovascular (CV) death (in the full population and in the population of patients with TSAT<20%) and reduce the rate of recurrent events of heart failure hospitalisations.

I.v. iron administration in the form of ferric carboxymaltosis (FCM) will be carried out according to the Summary of Product Characteristics (SmPC). Bolus administration (1000 mg) will be followed by an optional administration of 500-1000 mg within the first 4 weeks (up to a total of 2000 mg which is in-label) according to approved dosing rules, followed by administration of 500 mg FCM at every 4 months, except when haemoglobin is > 16.0 g/dL or ferritin is > 800 µg/L.

In the verum group, all patients will receive a saline administration, when no iron is indicated at the time of the visit and according to the values listed above. Patients originally assigned to the placebo group will receive a saline administration at all visits.

In the control group i.v. NaCl at a volume according to the dosing rules for FCM at all visits will be administered in a double-blind manner.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic HFrEF (CHF) of at least 3 months duration and a history of documented LVEF<45%.
2. Confirmed presence of ID (ferritin < 100 ng/mL or ferritin 100 - 299 ng/mL with TSAT < 20 %)
3. Serum haemoglobin of 9.5 - 14.0 g/dL
4. At time of screening considered re-stabilised and planned for discharge within next 24 h (NYHA 2 or 3), or stable ambulatory with a HF hospitalisation in the past 12 months (NYHA 2-4), or stable ambulatory with BNP > 100 pg/mL or NT-proBNP > 300 pg/mL or MR-proANP > 120 pmol/L (NYHA 2-4)
5. Written informed consent

Exclusion Criteria:

1. Hypersensitivity to the active substance, to FCM or any of its excipients
2. Known serious hypersensitivity to other parenteral iron products
3. Anaemia not attributed to iron deficiency, e.g. other microcytic anaemia
4. Evidence of iron overload or disturbances in the utilisation of iron
5. History of severe asthma with known FEV1 <50%
6. Acute bacterial infection
7. Presence of a deficiency for vitamin B12 and/or serum folate (if present, this needs to be corrected first)
8. Use of renal replacement therapy
9. Treatment with an erythropoietin stimulating agent (ESA), any i.v. iron and/or a blood transfusion in the previous 6 weeks prior to randomisation.
10. More than 500 meters in the initial 6-minutes walking-test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1105 (Actual)
Dates: Start 2017-03-07 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Time-to-first event of CV death or HF hospitalisation | The whole follow-up period. We aim for a minimum average follow-up of >2 years. We aim for a minimum follow-up of 6 months for all patients, but not less than 3 months.
  Show that treatment of patients with systolic heart failure (HF) and iron deficiency (ID) with i.v. iron (Ferric Carboxymaltose, FCM) versus placebo (i.v. NaCl) can extend the time-to-first-event of heart failure hospitalisations and cardiovascular (CV) death.
  Type I error rate control across the three primary endpoints will be ensured by using the Hochberg procedure.
Rate of total (first and recurrent) events of hospitalisations for heart failure (HF) | The wohle follow-up period. We aim for a minimum average follow-up of >2 years. We aim for a minimum follow-up of 6 months for all patients, but not less than 3 months.
  Show that treatment of patients with systolic heart failure (HF) and iron deficiency (ID) with i.v. iron (Ferric Carboxymaltose, FCM) versus placebo (i.v. NaCl) reduces the rate of recurrent events of heart failure hospitalisations.
Time-to-first event of CV death or HF hospitalisation in patients with TSAT <20% | During the wohle follow-up period. We aim for a minimum average follow-up of >2 years. We aim for a minimum follow-up of 6 months for all patients, but not less than 3 months.
  Show that treatment of patients with systolic heart failure (HF) and iron deficiency (ID) with i.v. iron (Ferric Carboxymaltose, FCM) versus placebo (i.v. NaCl) can extend the time-to-first-event of heart failure hospitalisations and cardiovascular (CV) death in the population of patients with TSAT<20%.

SECONDARY OUTCOMES:
Changes in 6-minute walk-test (nomogram) | The wohle follow-up period. We aim for a minimum average follow-up of >2 years. We aim for a minimum follow-up of 6 months for all patients, but not less than 3 months.
  Changes in 6-minute walk-test during follow-up
Changes in NYHA (New York Heart Association) functional class (scale) | The wohle follow-up period. We aim for a minimum average follow-up of >2 years. We aim for a minimum follow-up of 6 months for all patients, but not less than 3 months.
  Changes in NYHA functional class during follow-up
Changes in EQ-5D (questionnaire) | The wohle follow-up period. We aim for a minimum average follow-up of >2 years. We aim for a minimum follow-up of 6 months for all patients, but not less than 3 months.
  Changes EQ-5D during follow-up
Changes in Patient Global Assessment (PGA) of wellbeing (questionnaire) | The wohle follow-up period. We aim for a minimum average follow-up of >2 years. We aim for a minimum follow-up of 6 months for all patients, but not less than 3 months.
  Changes in PGA of wellbeing during follow-up
Changes in renal parameters (laboratory parameters) | The wohle follow-up period. We aim for a minimum average follow-up of >2 years. We aim for a minimum follow-up of 6 months for all patients, but not less than 3 months.
  Changes in renal parameters from baseline to end of follow-up, assessing creatinine levels
Changes in cardiovascular parameters (laboratory parameters) | The wohle follow-up period. We aim for a minimum average follow-up of >2 years. We aim for a minimum follow-up of 6 months for all patients, but not less than 3 months.
  Changes in cardiovascular parameters from baseline to end of follow-up, assessing natriuretic peptide levels
Changes in inflammatory parameters (laboratory parameters) | The wohle follow-up period. We aim for a minimum average follow-up of >2 years. We aim for a minimum follow-up of 6 months for all patients, but not less than 3 months.
  Changes in inflammatory parameters from baseline to end of follow-up, assessing C-reactive protein levels
Changes in metabolic parameters (laboratory parameters) | The wohle follow-up period. We aim for a minimum average follow-up of >2 years. We aim for a minimum follow-up of 6 months for all patients, but not less than 3 months.
  Changes in metabolic parameters from baseline to end of follow-up, assessing aspartate or alanine transaminase levels
Key Safety Endpoint: cardiovascular mortality | 36 months of follow-up
  cardiovascular mortality during 36 months of follow-up
Key Safety Endpoint: All-cause mortality | 36 months of follow-up
  All-cause mortality during 36 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Mahir Karaks, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (51):
- Germany (29):
  - Cardiologicum Hamburg, Hamburg, Hamburg
  - SLK-Kliniken Heilbronn GmbH Klinikum am Plattenwald, Bad Friedrichshall
  - Kerckhoff Klinik Bad Nauheim, Bad Nauheim
  - Universitätsmedizin Berlin Campus Benjamin Franklin, Berlin
  - Charité Berlin (Campus Virchow-Klinikum), Berlin
  - Stiftung Bremer Herzen Bremer Institut für Herz- und Kreislauf- Forschung, Bremen
  - Herzzentrum Dresden, Universitätsklinik, Dresden
  - Universitätsmedizin Göttingen, Göttingen
  - Uniklinik Greifswald, Klinik und Poliklinik für Innere Medizin B, Greifswald
  - Universitätsklinikum Halle (Saale), Halle
  - Universitärsklinikum Hamburg-Eppendorf, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Jena, Kardiologie, Jena
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Universitätsklinikum Schleswig-Holstein Campus Lübeck, Lübeck
  - Universitätsklinikum Magdeburg, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsmedizin Mannheim, Mannheim
  - Kliniken Maria Hilf GmbH, Innere Medizin II, Klinik für Kardiologie, Mönchengladbach
  - Praxis Dr. Schön Mühldorf, Mühldorf
  - LMU München Medizinische Klinik und Poliklinik 1, München
  - Klinikum rechts der Isar I. Medizinische Klinik und Poliklinik, München
  - Gemeinschaftspraxis Hagenmiller/ Jeserich, Nuremberg
  - Universitätsklinik Medizinische Klinik 8 - Kardiologie Paracelsus Medizinische Privatuniversität Klinikum Nürnberg, Campus Süd, Nuremberg
  - KardioPrax Remscheid, Remscheid
  - Kardiologische Praxis Dr. Jens Placke, Rostock
  - Studienzentrum Herzklinik Ulm GbR, Ulm
  - Universitätsklinikum Ulm, Ulm
- Hungary (6):
  - Szent Imre Kórház, Budapest
  - Semmelweis Egyetem, Budapest
  - Szent János kórház és Észak-budai Egyesített kórházak, Budapest
  - Honvéd Kórház, Budapest
  - Almási Balogh Pál Kórház, Ózd
  - Pécsi Orvostudományi, Pécs
- IRCCS San Raffaele Pisana (06-01), Rome, Italy
- Poland (5):
  - Cermed Hernik (05-07), Bialystok
  - Oddział Kardiologii Uniwersyteckiego (05-06), Opole
  - Klinika Niewydolności Serca I Transplantologii (05-04), Warsaw
  - Wroclaw Medical University (05-01), Warsaw
  - KLIMED Marek Klimkiewicz Lomza (05-05), Łomża
- Portugal (2):
  - Hospital de la Luz, Lisbon
  - Santa Maria University Hospital, Lisbon
- Slovenia (3):
  - University Medical Centre Ljubljana (07-03), Ljubljana
  - General Hospital Murska Sobota Division of Cardiology (07-01), Murska Sobota
  - Hospital Topolšica (07-03), Topolšica
- Spain (5):
  - Hospital del Mar (04-01), Barcelona
  - Hospital Universitario Clinico San Carlos Madrid (04-04), Madrid
  - Hospital Universitarion Virgen de la Victoria (04-03), Málaga
  - Hospital Clinico Universitario Valencia (04-02), Valencia
  - Hospital la Fe de Valencia (04-05), Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karakas M, Friede T, Butler J, Talha KM, Placzek M, Asendorf T, Diek M, Nosko A, Stas A, Kluge S, Jarczak D, DeHeer G, Rybczynski M, Bayes-Genis A, Bohm M, Coats AJS, Edelmann F, Filippatos G, Hasenfuss G, Haverkamp W, Lainscak M, Landmesser U, Macdougall IC, Merkely B, Pieske BM, Pinto FJ, Rassaf T, Visser-Rogers JK, Rosano G, Volterrani M, von Haehling S, Anker MS, Doehner W, Ince H, Koehler F, Savarese G, Khan MS, Krohnert UR, Gori T, Trenkwalder T, Akin I, Paitazoglou C, Kobielusz-Gembala I, Kuthi L, Frey N, Licka M, Kaab S, Laugwitz KL, Ponikowski P, Anker SD. Intravenous ferric carboxymaltose in heart failure with iron deficiency (FAIR-HF2 DZHK05 trial): Sex-specific outcomes. Eur J Heart Fail. 2025 Nov;27(11):2328-2342. doi: 10.1002/ejhf.3742. Epub 2025 Jul 31. PMID 40740027
- [Derived] Anker SD, Friede T, Butler J, Talha KM, Placzek M, Diek M, Nosko A, Stas A, Kluge S, Jarczak D, Deheer G, Rybczynski M, Bayes-Genis A, Edelmann F, Filippatos G, Hasenfuss G, Haverkamp W, Lainscak M, Landmesser U, Macdougall IC, Merkely B, Pieske BM, Pinto FJ, Rassaf T, Volterrani M, von Haehling S, Anker MS, Doehner W, Ince H, Koehler F, Savarese G, Rauch-Krohnert U, Gori T, Trenkwalder T, Akin I, Paitazoglou C, Kobielusz-Gembala I, Zmuda W, Kuthi L, Frey N, Licka M, Kaab S, Laugwitz KL, Ponikowski P, Karakas M. Ferric carboxymaltose assessment of morbidity and mortality in patients with iron deficiency and chronic heart failure (FAIR-HF2-DZHK05) trial: Baseline characteristics and comparison to other relevant clinical trials. Eur J Heart Fail. 2025 Aug;27(8):1436-1443. doi: 10.1002/ejhf.3658. Epub 2025 Apr 29. PMID 40300786
- [Derived] Anker SD, Friede T, Butler J, Talha KM, Placzek M, Diek M, Nosko A, Stas A, Kluge S, Jarczak D, deHeer G, Rybczynski M, Bayes-Genis A, Bohm M, Coats AJS, Edelmann F, Filippatos G, Hasenfuss G, Haverkamp W, Lainscak M, Landmesser U, Macdougall IC, Merkely B, Pieske BM, Pinto FJ, Rassaf T, Visser-Rogers JK, Rosano G, Volterrani M, von Haehling S, Anker MS, Doehner W, Ince H, Koehler F, Savarese G, Khan MS, Rauch-Krohnert U, Gori T, Trenkwalder T, Akin I, Paitazoglou C, Kobielusz-Gembala I, Kuthi L, Frey N, Licka M, Kaab S, Laugwitz KL, Ponikowski P, Karakas M. Intravenous Ferric Carboxymaltose in Heart Failure With Iron Deficiency: The FAIR-HF2 DZHK05 Randomized Clinical Trial. JAMA. 2025 Jun 10;333(22):1965-1976. doi: 10.1001/jama.2025.3833. PMID 40159390